CLINICAL TRIAL: NCT01830205
Title: Single Dose Pharmacokinetics and Safety of Daclatasvir in Subjects With Renal Function Impairment
Brief Title: Pharmacokinetic and Safety Study of Daclatasvir in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-063
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Normal renal function): Daclatasvir (Experimental): Daclatasvir 60 mg tablet by mouth single dose on Day 1
  Interventions: Drug: Daclatasvir
- Group B (End Stage Renal Disease): Daclatasvir (Experimental): Daclatasvir 60 mg tablet by mouth single dose on Day 1
  Interventions: Drug: Daclatasvir
- Group C (Moderate renal impairment): Daclatasvir (Experimental): Daclatasvir 60 mg tablet by mouth single dose on Day 1
  Interventions: Drug: Daclatasvir
- Group D (Severe renal impairment): Daclatasvir (Experimental): Daclatasvir 60 mg tablet by mouth single dose on Day 1
  Interventions: Drug: Daclatasvir

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052

SUMMARY:
The purpose of this study is to assess the effect of renal function impairment on the single dose pharmacokinetics of Daclatasvir.

DETAILED DESCRIPTION:
Treatment, Parallel Assignment, Open Label, Non-Randomized, Single Dose Adaptive Design, Pharmacokinetics Study

ELIGIBILITY:
Inclusion Criteria:

- Meet renal function criteria in one of four categories

Exclusion Criteria:

- Unstable or uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Davita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- [Derived] Garimella T, Wang R, Luo WL, Hwang C, Sherman D, Kandoussi H, Marbury TC, Alcorn H, Bertz R, Bifano M. Single-dose pharmacokinetics and safety of daclatasvir in subjects with renal function impairment. Antivir Ther. 2015;20(5):535-43. doi: 10.3851/IMP2941. Epub 2015 Feb 5. PMID 25654812
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 centers in United States of America.
Pre-assignment Details: A total of 58 participants were enrolled and 36 were treated with study drug. Remaining 22 were not treated (14 no longer met study criteria, 4 other reasons, 2 administrative reasons and 2 withdrew consent). Participants were grouped by Cockcroft-Gault creatine clearance method for primary analysis.
Groups:
- Normal Renal Function/Mild Renal Impairment: Participants with normal renal function and had creatinine clearance by the Cockcroft-Gault method >=90 milliliter per minute were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. One participant from this group, who had estimated glomerular filtration rate (eGFR) 60-89 mL/min per 1.73 m^2, was reallocated into mild renal impairment reporting arm and was administered with a single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. Original allocation was based on an estimated eGFR, while the reallocation was based on the eGFR measurement at baseline.
- Mild/Moderate Renal Impairment: Participants with moderate renal impairment and had eGFR 30-59 mL/min per 1.73 m^2 were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. Two participants from this group, who had eGFR 60-89 mL/min per 1.73 m^2, were reallocated into mild renal impairment reporting arm and were administered with a single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. Original allocation was based on an estimated eGFR, while the reallocation was based on the eGFR measurement at baseline.
- Mild/Severe Renal Impairment: Participants with severe renal impairment and had eGFR 15 to 29 mL/min per 1.73 m^2 were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. One participant from this group, who had eGFR 60-89 mL/min per 1.73 m^2, was reallocated into mild renal impairment reporting arm and was administered with a single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. Original allocation was based on an estimated eGFR, while the reallocation was based on the eGFR measurement at baseline.
- End Stage Renal Disease: Participants with end stage renal disease and had eGFR <15 mL/ min per 1.73 m^2, with or without hemodialysis were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
Period: Overall Study
Arm/Group | Normal Renal Function/Mild Renal Impairment | Mild/Moderate Renal Impairment | Mild/Severe Renal Impairment | End Stage Renal Disease
Started | 12 | 6 | 6 | 12
Completed | 12 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Renal Function/Mild Renal Impairment: Participants with normal renal function and had creatinine clearance by the Cockcroft-Gault method >=90 milliliter per minute were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. One participant from this group, who had eGFR 60-89 mL/min per 1.73 m^2, was reallocated into mild renal impairment reporting arm and was administered with a single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. Original allocation was based on an estimated eGFR, while the reallocation was based on the eGFR measurement at baseline.
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function/Mild Renal Impairment | Mild/Moderate Renal Impairment | Mild/Severe Renal Impairment | End Stage Renal Disease | Total
Number analyzed (Participants) | 12 | 6 | 6 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (8.5) | 62.0 (12.6) | 66.3 (9.9) | 49.0 (11.7) | 53.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 6
  Male | 11 | 4 | 4 | 11 | 30
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 6 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(INF)] of Daclatasvir
Description: AUC(INF) was estimated by summing the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration and the extrapolated area, computed by the quotient of the last observable concentration and elimination rate constant. The pharmacokinetic (PK) analysis was based on Cockcroft-Gault (C-G) creatinine clearance (CLcr) grouping method: normal renal function, end stage renal disease (ESRD), moderate and severe renal impairment. Mild participants were counted as per their original allocation.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: PK data set included all participants who received at least 1 dose of daclatasvir with adequate PK profiles. The PK analysis was based on the C-G CLcr grouping method: normal renal function (n=11), ESRD (n=10), moderate (n=5) and severe renal impairment (n=6). Mild participants (n=4) are also counted as per their original allocation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*h/mL)
Groups:
- Normal Renal Function: Participants with normal renal function and had creatinine clearance by the Cockcroft-Gault method >= 90 milliliter per minute were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
- Mild Renal Impairment: Participants were reallocated from other arms (normal, moderate and severe renal impairment) with mild renal impairment who had eGFR 60-89 mL/min per 1.73 m^2 were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
- Moderate Renal Impairment: Participants with moderate renal impairment and had eGFR 30-59 mL/min per 1.73 m^2 were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
- Severe Renal Impairment: Participants with severe renal impairment and had eGFR 15 to 29 mL/min per 1.73 m^2 were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
- End Stage Renal Disease: Participants with end stage renal disease and had estimated glomerular filtration rate (eGFR) < 15 mL/ min per 1.73 m^2, with or without hemodialysis were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
nanograms*hours/milliliter (ng*h/mL) | 11215.264 (40) | 21261.199 (62) | 24789.951 (35) | 21946.450 (39) | 14257.489 (25)

2. Secondary Outcome: Unbound Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity Time (AUC(INF)u) of Daclatasvir
Description: AUC(INF)u was calculated by multiplying the area under the plasma concentration-time curve from time zero extrapolated to infinite time by mean fraction of unbound drug from 1 hour post-dose time point.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: Pharmacokinetic (PK) data set included all participants who received at least 1 dose of daclatasvir with adequate PK profiles. The PK analysis was based on C-G CLcr grouping method: normal renal function (n=11), ESRD (n=10), moderate (n=5) and severe renal impairment (n=6). Mild participants (n=4) are also counted as per their original allocation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- End Stage Renal Disease: Participants with end stage renal disease and had estimated glomerular filtration rate (eGFR) <15 mL/ min per 1.73 m^2, with or without hemodialysis were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
ng*h/mL | 83.845 (37) | 128.157 (41) | 144.915 (13) | 139.576 (43) | 100.736 (31)

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Daclatasvir
Description: Maximum observed plasma concentration following drug administration from the raw plasma concentration-time data. The plasma samples were analyzed for daclatasvir by using a validated liquid chromatography tandem mass spectrometric (LC-MS/MS) assay.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
ng/mL | 1111.497 (39) | 1619.572 (13) | 1745.845 (31) | 1207.137 (33) | 1085.344 (15)

4. Secondary Outcome: Unbound Maximum Observed Plasma Concentrations of Daclatasvir
Description: Unbound Maximum observed plasma concentrations (Cmaxu) was calculated by multiplying maximum observed plasma concentrations by mean fraction of unbound drug from 1 hour post-dose time point.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
ng/mL | 8.309 (34) | 9.762 (14) | 10.206 (20) | 7.677 (33) | 7.668 (36)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Last Measurable Concentration [AUC(0-T)] of Daclatasvir
Description: AUC(0-T) was calculated as the sum of linear trapezoids using non-compartmental analysis.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: Pharmacokinetic (PK) data set included all participants who received at least 1 dose of daclatasvir with adequate PK profiles. The analysis was based on C-G CLcr grouping method: normal renal function (n=11), ESRD (n=10), moderate (n=5) and severe renal impairment (n=6). Mild participants (n=4) are also counted as per their original allocation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour (h)/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
ng*hour (h)/mL | 11092.967 (40) | 20852.129 (60) | 24343.711 (36) | 21238.909 (37) | 13934.562 (25)

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Daclatasvir
Description: Tmax was defined as the time required to reach maximum observed plasma concentration. Tmax was directly determined from the raw plasma concentration-time data.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
hours | 1.000 [1.00 to 2.00] | 1.250 [1.00 to 1.50] | 1.000 [1.00 to 2.00] | 1.500 [1.00 to 3.00] | 1.250 [1.00 to 4.00]

7. Secondary Outcome: Plasma Half-life (T-half) of Daclatasvir
Description: Terminal half-life was the time required for one half of the total amount of administered drug eliminated from the body.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
hours | 13.625 (25) | 15.661 (31) | 16.912 (19) | 20.224 (24) | 15.678 (37)

8. Secondary Outcome: Apparent Total Body Clearance (CLT/F) of Daclatasvir
Description: Apparent total body clearance was calculated by dividing the dose by area under the plasma concentration-time curve from time zero extrapolated to infinite time.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/minute (mL/min)
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
milliliter/minute (mL/min) | 89.164 (26) | 47.034 (43) | 40.339 (27) | 45.565 (31) | 70.139 (33)

9. Secondary Outcome: Unbound Apparent Clearance (CLU/F) of Daclatasvir
Description: The CLU/F was calculated by dividing the apparent total body clearance by mean fraction of unbound drug from 1 hour post dose time point.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
mL/min | 11926.796 (53) | 7802.955 (33) | 6900.602 (13) | 7164.575 (41) | 9926.962 (35)

10. Secondary Outcome: Percent Urinary Recovery (%UR) of Daclatasvir
Description: The percentage of daclatasvir recovered in the urine was determined by using validated liquid chromatography-tandem mass spectrometry methods. The sum of the percentage of dose recovered in urine from all intervals was calculated to obtain the total percentage of urinary excretion.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: Pharmacokinetic (PK) data set included all participants who received at least 1 dose of daclatasvir with adequate PK profiles. The PK analysis was based on C-G CLcr grouping method: normal renal function (n=11), ESRD (n=3), moderate (n=5) and severe renal impairment (n=5). Mild participants (n=4) are also counted as per their original allocation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of daclatasvir recovered
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 5 | 3
Percentage of daclatasvir recovered | 5.007 (36) | 5.820 (27) | 3.530 (40) | 2.658 (58) | 0.199 (131)

11. Secondary Outcome: Renal Clearance (CLR) of Daclatasvir
Description: The CLR was calculated by dividing the total amount excreted in the urine from 0 to 96 hours by the area under the plasma concentration-time curve from time zero extrapolated to infinite time.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 5 | 3
mL/min | 4.465 (29) | 2.737 (28) | 1.424 (48) | 1.165 (37) | 0.147 (114)

12. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Daclatasvir
Description: The Vd/F was calculated by dividing the product of the dose and mean residence time by area under the plasma concentration-time curve from time zero extrapolated to infinite time.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- Mild Renal Impairment: Participants were re-randomized from other arms (normal, moderate and severe renal impairment) with mild renal impairment who had eGFR 60-89 mL/min per 1.73 m^2 were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 11 | 4 | 5 | 6 | 10
Liters | 105.157 (37) | 63.761 (30) | 59.054 (36) | 79.769 (35) | 95.186 (37)

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events and Who Died
Description: Adverse event (AE) was defined as any new unfavorable symptom, sign, or disease or worsening of a pre-existing condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalisation.
Time Frame: First dose up to Day 5 post last dose for AEs; up to 30 days post last dose for SAEs
Population: Analysis was done in safety data set population, defined as all the participants who received the study medication.
Measure: Number; unit: Participants
Groups:
- Mild/Moderate Renal Impairment: Participants with moderate renal impairment and had eGFR 30-59 mL/min per 1.73 m^2 were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. Two participants from this group, who had eGFR 60-89 mL/min per 1.73 m^2, were reallocated into mild renal impairment reporting arm and were administered with a single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1.Original allocation was based on an estimated eGFR, while the reallocation was based on the eGFR measurement at baseline.
Arm/Group | Normal Renal Function/Mild Renal Impairment | Mild/Moderate Renal Impairment | Mild/Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 12 | 6 | 6 | 12
Participants
  SAEs | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0
  Discontinuations due to AEs | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Marked Abnormalities Reported as Adverse Events
Description: Significant laboratory abnormalities were defined as any test results which were observed beyond the clinically acceptable limits as per the discretion of investigator.
Time Frame: Baseline up to Day 5 post dose
Population: The analysis was done in safety population.
Measure: Number; unit: Participants
Arm/Group | Normal Renal Function/Mild Renal Impairment | Mild/Moderate Renal Impairment | Mild/Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 12 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Electrocardiogram (ECG) Reported as Adverse Events
Description: The number of participants with clinically relevant changes in ECG which were considered as adverse events was determined.
Time Frame: Baseline up to Day 5 post dose
Population: Analysis was done in safety data set population.
Measure: Number; unit: Participants
Arm/Group | Normal Renal Function/Mild Renal Impairment | Mild/Moderate Renal Impairment | Mild/Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 12 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Out-of-range Vital Signs Reported as Adverse Events
Description: The total number of participants with abnormal range vital signs which were considered as adverse events was determined.
Time Frame: Baseline up to Day 5 post dose
Population: Analysis was done in safety data set population.
Measure: Number; unit: Participants
Arm/Group | Normal Renal Function/Mild Renal Impairment | Mild/Moderate Renal Impairment | Mild/Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 12 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: First dose up to Day 5 post last dose of study treatment for AEs; up to 30 days post last dose for SAEs
Groups:
- Group-A: Participants with normal renal function and had creatinine clearance by the Cockcroft-Gault method >=90 milliliter per minute were administered with single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. One participant from this group, who had eGFR 60-89 mL/min per 1.73 m^2, was reallocated into mild renal impairment reporting arm and was administered with a single oral dose of daclatasvir 60 mg tablet after 10 hours of overnight fasting on Day 1. Original allocation was based on an estimated eGFR, while the reallocation was based on the eGFR measurement at baseline.
Arm/Group | Group-A | Mild/Moderate Renal Impairment | Mild/Severe Renal Impairment | End Stage Renal Disease
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/6 | 1/6 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group-A (N=12) | Mild/Moderate Renal Impairment (N=6) | Mild/Severe Renal Impairment (N=6) | End Stage Renal Disease (N=12)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.